CLINICAL TRIAL: NCT06296953
Title: Safety and Feasibility of the PERIsign System in Demonstrating Involuntary Muscle Defense as a Sign of Peritonitis in Subjects With Appendicitis
Brief Title: Safety & Feasibility of PERIsign System in Demonstrating Involuntary Muscle Defense as a Sign of Peritonitis in Subjects With Appendicitis
Acronym: PeriSaFe01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: STB INN AB (Industry)
Collaborators: Aurevia (Industry); Region Halland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PeriSaFe01; CIV-23-11-044875 (Other: Swedish Medical Product Agency)
Record Dates: First submitted 2024-02-10; First posted 2024-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Appendicitis Acute; Appendicitis; Abdominal Pain; Peritonitis
Keywords: Appendicitis; Acute abdominal pain; Peritonitis; Medical Device; PERIsign
MeSH Terms: conditions — Appendicitis; Abdominal Pain; Peritonitis; Abdomen, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Group (Experimental): Patient will be examined with the new device, PERIsign.
  Interventions: Device: PERIsign examination
- Healthy Volunteers (Active Comparator): The group will also be examined with the device, PERIsign
  Interventions: Device: PERIsign examination

INTERVENTIONS:
Device: PERIsign examination — Patients will be examined with the new device, PERIsign

SUMMARY:
This will be an explorative, proof-of-principle, open, multi-center investigation.

The investigation aims to investigate the safety of the PERIsign system and the ability of physicians to differentiate between healthy individuals and subjects with involuntary muscle defense as a sign of peritonitis by utilizing PERIsign data. The investigation will include a total of 20 subjects admitted to hospital for suspected appendicitis and planned for emergency surgery and 20 healthy volunteers. Both male and female subjects aged 18-70 years will be enrolled.

All subjects will undergo PERIsign examinations. Subjects with suspected appendicitis will undergo 1-2 PERIsign examinations before their planned appendectomy surgery. For the healthy volunteers, there is only 1 PERIsign examination. During each examination, 4 PERIsign curves will be obtained, one from each quadrant of the abdomen. The attending physician will interpret the appearance of the PERIsign curves of all subjects, including those from the healthy volunteers. The duration of the PERIsign examination will be documented, and usability data will be gathered, including the need for sensor adjustments, subject perception of the examination, and any discomfort experienced. In addition, blinded physicians will evaluate all subjects' PERIsign curves and determine whether each subject has involuntary muscle defense as a sign of peritonitis. These blinded physicians will have access to all 4 PERIsign curves obtained during each examination, while other data will not be disclosed to them.

Safety will be evaluated through analysis of reported adverse events and device deficiencies

DETAILED DESCRIPTION:
METHODOLOGY The PERIsign system is intended to aid physicians in demonstrating involuntary muscle defense as a sign of peritonitis by assessing involuntary activity in abdominal muscles by use of sEMG sensors and induced pressure.

In this investigation, all subjects will undergo examinations with the PERIsign system. For subjects with suspected appendicitis, assessments will be performed at the clinic on up to 2 occasions. An initial examination will occur when the patient is scheduled for surgery and admitted to the hospital. The following examination is optional and will occur 4-6 hours after the initial examination but before their planned surgery. Post-operative clinical assessments, patho-anatomical diagnosis and clinical end diagnosis will be collected from medical journals, 30 ±5 days after the initial examination. For the healthy volunteers, there is only 1 examination.

INVESTIGATIONAL MEDICAL DEVICE The PERIsign system is a medical device designed to measure the contractions of the internus and externus oblique muscles in the abdomen by use of surface electromyography (sEMG) sensors and induced pressure to facilitate the evaluation of a patient with acute abdominal pain. The PERIsign system aims to aid physicians in demonstrating involuntary muscle defense as a sign of peritonitis, an inflammation of the peritoneum, by measuring muscle activity both at rest and in response to pressure on the abdominal wall.

The PERIsign Minimal Viable Product is the first iteration of the device and will be used for the present clinical investigation. It comprises four sensor heads with connections, used together with single use sensor electrodes, that are applied to four specific locations on the patient's abdomen, and one reference electrode attached to the hand. Each sensor head has a pressure sensor on top that measures the pressure applied to the sensor, mimicking the manual palpation performed by a physician. The PERIsign system will display and record the patient's muscle activity and the pressure being applied to their abdomen. PERIsign is connected to a laptop for data collection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy volunteers

For enrolment in the investigation, healthy volunteers must fulfil all the following criteria:

1. Subject is 18-70 years of age
2. The subject reports having understood and has signed the Informed Consent Form (ICF) and is willing to comply with all assessments
3. The subject should have a sufficient height and physical build to enable the attachment of the PERIsign sensors to their abdomen, as judged by the Investigator Inclusion criteria for the patient group

For enrolment in the investigation, patients must fulfil all the following criteria:

1. Patient is 18-70 years of age
2. The patient reports having understood and has signed the ICF and is willing to comply with all assessments
3. The patient is admitted to the hospital with suspected appendicitis and scheduled for emergency surgery within 24 hours.
4. Patient is deemed clinically stable, as judged by the Investigator
5. The patient should have a sufficient height and physical build to enable the attachment of the PERIsign sensors to their abdomen, as judged by the Investigator

Exclusion Criteria:

Exclusion criteria for healthy volunteers

Healthy volunteers meeting any of the following criteria will not be permitted to enter the investigation:

1. BMI >30
2. Presence of any known pathological diseases in the abdomen
3. Subject who previously underwent abdominal surgery
4. Subject with spinal cord injury
5. Subject with pacemaker
6. Pregnancy at the time of enrollment, as confirmed by either knowledge or a urine test
7. The subject has a cognitive incapacity or language barrier precluding adequate understanding or cooperation
8. The subject is considered by the Investigator to be unsuitable to participate in the investigation for any other reason
9. Subject already enrolled (within 30 days prior to enrolment) in another investigational drug/s or device/s clinical study Exclusion criteria for the patient group

Patients meeting any of the following criteria will not be permitted to enter the investigation:

1. BMI >30
2. Patient who previously underwent abdominal surgery
3. The patient is currently undergoing immunosuppressive therapy, including systemic corticosteroid treatment for two weeks prior to enrollment
4. Patient with spinal cord injury
5. Patient with pacemaker
6. Known abdominal ventral hernia
7. Known abdominal rectus muscle diastasis
8. Retrocecal appendix according to radiology
9. Other known pathological conditions of the abdomen that may interfere with the performance, evaluation and outcome of the clinical evaluation, as determined by the Investigator
10. The patient must not be pregnant at the time of enrollment, as confirmed by either prior knowledge or a urine test
11. The patient has a cognitive incapacity or language barrier precluding adequate understanding or cooperation
12. The patient is considered by the Investigator to be unsuitable to participate in the investigation for any other reason
13. The PERIsign examination is deemed to interfere with the standard of care
14. Subject already enrolled (within 30 days prior to enrolment) in another investigational drug/s or device/s clinical study -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects experiencing any adverse events during the examination | 1 hour
  Evaluation of there is any adverse events during the examination of the new diagnostic device.
Proportion of device deficiencies during the evaluation | 1 hour
  Evaluation of there is any device deficiencies during the examination of the new diagnostic device.

SECONDARY OUTCOMES:
To estimate the sensitivity and specificity of diagnosing pathological muscle defense when using the PERIsign system | 1 hour
  During the evaluation the examiner interprets the graphical curves presented by the PERIsign system to evaluate and determine if there is an involuntary muscle defense at the subjects abdominal wall. The sensitivity and specificity will be calculated.
Proportion of examinations of the PERIsign system that its performed without usability issues. | 1 hour
  The usability of the PERIsign system is tested by measuring how long the examination will take and how easy it is to use bye the examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lindskog, ass. Prof, Principal Investigator — Region Halland
Locations (2):
- Sweden (2):
  - Hallands Sjukhus Halmstad, Halmstad
  - Hallands Sjukhus Varberg, Varberg

IPD SHARING:
Plan to Share IPD: No